CLINICAL TRIAL: NCT02971683
Title: A Phase 3, Randomized, Double-Blind Clinical Trial to Evaluate the Efficacy and Safety of Abatacept SC With Standard Treatment Compared to Standard Treatment Alone in Improving Disease Activity in Adults With Active Idiopathic Inflammatory Myopathy (IIM)
Brief Title: Trial to Evaluate the Efficacy and Safety of Abatacept in Combination With Standard Therapy Compared to Standard Therapy Alone in Improving Disease Activity in Adults With Active Idiopathic Inflammatory Myopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM101-611; 2016-002269-77 (EudraCT Number)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Polymyositis; Dermatomyositis; Autoimmune Necrotizing Myopathy; Overlap Myositis; Juvenile Myositis Above the Age of 18
MeSH Terms: conditions — Polymyositis; Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abatacept subcutaneous + Standard Treatment (Active Comparator): Abatacept subcutaneous weekly in addition to the subject's current standard treatment for 24 weeks followed by a 28 week open-label period of abatacept treatment plus the subject's current standard treatment.
  Interventions: Drug: Abatacept subcutaneous
- Placebo of Abatacept subcutaneous + Standard Treatment (Placebo Comparator): Placebo of Abatacept subcutaneous weekly in addition to the subject's current standard treatment for 24 weeks followed by a 28 week open-label period of abatacept treatment plus the subject's current standard treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Abatacept subcutaneous — Specified dose of Abatacept subcutaneous on specified days
  Arms: Abatacept subcutaneous + Standard Treatment
Drug: Placebo — Placebo of Abatacept subcutaneous
  Arms: Placebo of Abatacept subcutaneous + Standard Treatment

SUMMARY:
Trial to Evaluate the Efficacy and Safety of Abatacept subcutaneous (SC) in Combination With Standard Therapy Compared to Standard Therapy Alone in Improving Disease Activity in Adults With Active Idiopathic Inflammatory Myopathy

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of IIM based on the Bohan and Peter classification criteria: i) Subjects with dermatomyositis (DM) must also have a confirmed myositis-associated rash (Gottron's papules or a heliotrope rash preferably confirmed by skin biopsy) and 2 or more of the remaining 4 criteria.

ii) Subjects with a diagnosis of IIM other than DM include PM, autoimmune necrotizing myopathy, myositis in association with another connective tissue disease (overlap myositis) and juvenile myositis subjects above the age of 18. These subjects must have a prior muscle biopsy diagnostic for IIM or a positive test for at least one myositis-specific autoantibody (anti-aminoacyl-tRNA synthetases (Jo-1, PL-7, PL-12, EJ, OJ, KS, Zo, YRS), anti-Mi-2, anti-SRP, anti-TIF1-g, anti-NXP-2, anti-MDA5, anti-SAE, anti-HMGCR). For subjects with overlap myositis, the myositis must be the principal clinically active manifestation of their disease. Where applicable, documentation of prior skin biopsy, muscle biopsy, and autoantibody results must be obtained and retained by the site.

* Demonstrable muscle weakness measured by the MMT-8 of ≤ 135 units and any 3 of the following: i) MMT-8 ≤ 125 units; ii) Physician's global assessment (PGA) visual analog scale (VAS) ≥2 cm; iii) Subject's global assessment (SGA) VAS ≥2 cm; iv) HAQ-DI ≥ 0.5; v) One or more muscle enzyme (CK, aldolase, LDH, AST, ALT) ³ 1.3 times upper limit of normal (ULN); vi) MDAAT Extramuscular Global Activity VAS ≥2 cm
* Demonstration of currently active IIM will be determined by an adjudication committee unless the subject has any one of the following: i) an active myositis-associated rash (Gottron's papules or heliotrope rash), or ii) a recent (within 3 months prior to signing informed consent) biopsy, magnetic resonance imaging (MRI), or electromyogram (EMG) demonstrating active disease, or iii) an elevated CK > 5 times the upper limit of normal
* Active disease despite prior treatment with corticosteroids, immunosuppressants, or biologics as determined by the investigator
* The subject must be on background standard treatment for IIM. The standard treatments that are allowed as background treatment for IIM includes: i) Corticosteroids alone, or ii) One of the following immunosuppressants: methotrexate, azathioprine, mycophenolate mofetil, tacrolimus, or cyclosporine (combinations of these treatments are not allowed), or iii) A combination of corticosteroids and one of the above immunosuppressants. The subject must have been on the same medication(s) for IIM for 12 weeks prior to randomization and the dose must have been stable for 4 weeks prior to randomization. If using azathioprine, the subject must have been on azathioprine for at least 24 weeks with a stable dose for at least 12 weeks prior to randomization.

Exclusion Criteria:

* Subjects with Inclusion Body Myositis (IBM), or myositis other than IIM, eg, drug-induced myositis and PM associated with HIV
* Subjects treated with penicillamine or zidovudine in the past 3 months
* Subjects treated with rituximab in the 6 months prior to randomization (there must be laboratory results indicating the presence of circulating B cells [CD19+]). Any other biologic treatment in the past 3 months or immune globulin (intravenous [IVIG] or subcutaneous [SCIG]) in the past 3 months prior to randomization
* Subjects with uncontrolled or rapidly progressive interstitial lung disease
* Subjects with severe muscle damage (Myositis Damage Index > 7/10), permanent weakness due to a non-IIM cause, or myositis with cardiac involvement
* Cancer-associated myositis (myositis diagnosed within 2 years of a diagnosis of cancer
* Subjects who are known to be positive for the anti-TIF-1 (p155/140) autoantibody prior to randomization who were diagnosed with IIM < 1 year prior to randomization.
* Subjects at risk for tuberculosis
* Subjects with recent acute infection requiring antibiotics
* Subjects with history of chronic or recurrent bacterial, viral or systemic fungal infections
* Subjects who have a present malignancy or have had a previous malignancy within the last 5 years prior to screening (except for a documented history of cured non-metastatic squamous or basal cell skin carcinoma or cervical carcinoma in situ).

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (79):
- United States (25):
  - Local Institution - 0015, Phoenix, Arizona
  - Local Institution - 0075, Beverly Hills, California
  - Local Institution - 0012, Orange, California
  - Local Institution - 0057, Washington D.C., District of Columbia
  - Local Institution - 0018, Fort Lauderdale, Florida
  - Local Institution - 0013, Miami, Florida
  - Local Institution - 0006, Kansas City, Kansas
  - Johns Hopkins University -Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Local Institution - 0058, Boston, Massachusetts
  - Local Institution - 0089, Ann Arbor, Michigan
  - Local Institution - 0002, Eagan, Minnesota
  - Local Institution - 0011, Omaha, Nebraska
  - Local Institution - 0004, Lebanon, New Hampshire
  - Local Institution - 0097, New York, New York
  - Local Institution - 0010, Wilmington, North Carolina
  - Local Institution - 0056, Columbus, Ohio
  - Local Institution - 0094, Middleburg Heights, Ohio
  - Local Institution - 0059, Norman, Oklahoma
  - Local Institution - 0055, Bethlehem, Pennsylvania
  - Local Institution - 0014, Pittsburgh, Pennsylvania
  - Local Institution - 0005, Orangeburg, South Carolina
  - Local Institution - 0017, Jackson, Tennessee
  - Local Institution - 0096, Austin, Texas
  - Local Institution - 0016, Houston, Texas
  - Local Institution - 0095, Seattle, Washington
- Australia (4):
  - Local Institution - 0051, Camperdown, New South Wales
  - Local Institution - 0053, St Leonards, New South Wales
  - Local Institution - 0035, Auchenflower, Queensland
  - Local Institution - 0036, Murdoch, Western Australia
- Brazil (7):
  - Local Institution - 0070, Vitória, Espírito Santo
  - Local Institution - 0073, Salvador, Estado de Bahia
  - Local Institution - 0069, Juiz de Fora, Minas Gerais
  - Local Institution - 0072, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0074, Bairro Jardim, São Paulo
  - Local Institution - 0067, Rio Grande
  - Local Institution - 0071, São Paulo
- Local Institution - 0029, Prague, Czechia
- France (5):
  - Local Institution - 0100, Brest
  - Local Institution - 0045, Clermont-Ferrand
  - Local Institution - 0043, Lille
  - Local Institution - 0042, Paris
  - Local Institution - 0044, Strasbourg
- Germany (4):
  - Local Institution - 0027, Berlin
  - Local Institution - 0054, Halle
  - Local Institution - 0028, Hamburg
  - Local Institution - 0030, München
- Italy (5):
  - Local Institution - 0023, Pavia, Lombardy
  - Local Institution - 0031, Ferrara
  - Local Institution - 0024, Florence
  - Local Institution - 0020, Padua
  - Local Institution - 0025, Pisa
- Japan (16):
  - Local Institution - 0091, Kitakyushu, Fukuoka
  - Local Institution - 0090, Sapporo, Hokkaido
  - Local Institution - 0078, Sapporo, Hokkaido
  - Local Institution - 0082, Tsukuba, Ibaraki
  - Local Institution - 0083, Kawasaki-shi, Kanagawa
  - Local Institution - 0084, Kumamoto, Kumamoto
  - Local Institution - 0088, Nagasaki, Nagasaki
  - Local Institution, Sasebo, Nagasaki
  - Local Institution - 0077, Iruma-gun, Saitama
  - Local Institution - 0086, Bunkyo-ku, Tokyo
  - Local Institution - 0079, Bunkyo-ku, Tokyo
  - Local Institution - 0081, Chuo-ku, Tokyo
  - Local Institution - 0092, Shinjuku-ku, Tokyo
  - Local Institution - 0093, Shinjuku-Ku, Tokyo
  - Local Institution - 0087, Ube-shi, Yamaguchi
  - Local Institution - 0076, Miyagi
- Mexico (5):
  - Local Institution - 0048, Guadalajara, Jalisco
  - Local Institution - 0049, Mexico City, Mexico City
  - Local Institution - 0046, Mexico City, Mexico City
  - Local Institution - 0047, San Luis Potosí City
  - Local Institution - 0052, San Luis Potosí City
- South Korea (3):
  - Local Institution - 0066, Seoul
  - Local Institution - 0065, Seoul
  - Local Institution - 0064, Seoul
- Sweden (4):
  - Local Institution - 0040, Lund
  - Local Institution - 0041, Örebro
  - Local Institution - 0037, Stockholm
  - Local Institution - 0038, Västerås

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept + Standard Treatment: Participants receive subcutaneous abatacept (125 mg weekly) in combination with standard treatment for the first 24 weeks (6 months) during the double-blind period. Participants continue to receive abatacept in the Open-Label and Long-Term Open Label Periods.
- Placebo + Standard Treatment: Participants receive placebo (to match subcutaneous abatacept) in combination with standard treatment for the first 24 weeks (6 months) during the double-blind period. Participants then switch from placebo to abatacept in the Open-Label and Long-Term Open Label Periods.
Period: Double-Blind (24 Weeks)
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Started (All participants who started the Double-Blind period were treated) | 75 | 73
Completed (Completed Period) | 69 | 65
Not Completed | 6 | 8
Not completed — Other reasons | 0 | 1
Not completed — Poor/Non-Compliance | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant withdrew consent | 1 | 1
Not completed — Participant request to discontinue study treatment | 1 | 1
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 2 | 2
Not completed — Participant no longer meets study criteria | 1 | 0
Period: Open-Label
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Started (All participants treated in the Open Label Period) | 69 | 63
Completed (Completed Period) | 65 | 61
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participants withdrew consent | 0 | 2
Not completed — Participant request to discontinue study treatment | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Period: Long-Term Open Label
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Started | 25 | 21
Completed (Completed Period) | 1 | 0
Not Completed | 24 | 21
Not completed — Administrative reason by sponsor | 20 | 17
Not completed — Participant withdrew consent | 1 | 0
Not completed — Participant request to discontinue study treatment | 1 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment | Total
Number analyzed (Participants) | 75 | 73 | 148
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (14.41) | 48.1 (14.09) | 48.7 (14.22)
Age, Customized [Number; unit: Participants]
  16-29 years old | 9 | 9 | 18
  30-39 years old | 8 | 14 | 22
  40-49 years old | 14 | 14 | 28
  50-59 years old | 31 | 19 | 50
  >/= 60 years old | 13 | 17 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 54 | 106
  Male | 23 | 19 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 49 | 51 | 100
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 10 | 6 | 16
  Black or African American | 9 | 8 | 17
  White | 42 | 42 | 84
  Japanese | 11 | 10 | 21
  Other | 0 | 3 | 3
  Unknown | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving International Myositis Assessment and Clinical Studies Definition of Improvement (IMACS DOI) at Week 24 Without Rescue
Description: The number of participants who achieve IMACS DOI (International Myositis Assessment and Clinical Studies definition of improvement) without rescue medication at week 24.
  The IMACS DOI is: An improvement of >/= 20% from baseline in 3 IMACS core measures, no more than 2 IMACS core measure scores worsen by >/= 25% from baseline, and no more than 2 IMACS core measure scores worsen by >/= 25% from baseline.
  IMACS core measures are: Physician Global Assessment of Disease Activity (PGA), Patient (Subject) Global Assessment of Disease Activity (SGA), Manual Muscle Test (MMT-8), Health Assessment Questionnaire-Disability Index (HAQ-DI), Muscle Enzyme levels, Myositis Disease Activity Assessment Tool (MDAAT) Extramuscular Global Activity.
Time Frame: From first dose to 24 weeks after first dose. (Approximately 169 days)
Population: All treated participants excluding participants with relevant protocol deviations
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 73
Participants | 42 [44.8 to 67.2] | 31 [31.6 to 54.5]
Statistical Analysis 1: Comparison: Abatacept + Standard Treatment; Test type: Superiority; p = 0.083, Regression, Logistic; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.9 to 3.5]

2. Secondary Outcome: Mean Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) From Baseline to Week 24
Description: The adjusted mean change from baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI). HAQ-DI is a patient-reported outcome measuring disability by asking a total of 20 questions in eight categories of function: dressing, arising, eating, walking, hygiene, reach, grip, and activities. If an aid or device is used or if help is required from another individual, then the minimum score for that section is 2. The highest component score in each category determines the score for the category and scores are averaged to give the disability index. The HAQ scale ranges from 0 (no difficulties) to 3 (unable to do).
Time Frame: From first dose to 24 weeks after first dose. (Approximately 169 days)
Population: All treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 66 | 62
Score on a scale | -0.31 (0.067) | -0.20 (0.069)

3. Secondary Outcome: Mean Change in Muscle Endurance Using the Myositis Function Index (FI-2) From Baseline to Week 24
Description: The adjusted mean change from baseline in Myositis FI-2 scores is assessing muscle endurance impairment by testing specific muscle groups. The 3 Score average includes shoulder flexion, hip flexion, and head lift. Each muscle group is scored as the number of correctly performed repetitions with 60 maximal number of repetitions.
  The total score is based on hip flexion, shoulder flexion (R/L) and neck divided by 3 (range 0-60 repetitions).
Time Frame: From first dose to 24 weeks after first dose. (Approximately 169 days)
Population: All treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: Number of repetitions
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 59 | 58
Number of repetitions | 4.1 (1.33) | 1.2 (1.38)

4. Secondary Outcome: Mean Change in Myositis Disease Activity Assessment Tool (MDAAT) Assessment of Extra-muscular From Baseline to Week 24
Description: The adjusted mean change from baseline in the Myositis Disease Activity Assessment Tool (MDAAT) assessment of extra-muscular uses a 100 mm Visual Analog Scale (VAS) scale. This VAS assesses the overall extra-muscular clinical features based upon: 1) The presence of clinical features or symptoms within the previous 4 weeks that are due to active disease. 2) The judgment that the feature is due to the myositis disease process. 3) The concept that disease activity is defined as a potentially reversible finding. 4) A clinical, functional, and laboratory assessments.
  The scoring is performed by the investigator and ranges from 0 (absent extra-muscular disease activity) to 100 (maximum extra-muscular disease activity).
Time Frame: From first dose to 24 weeks after first dose. (Approximately 169 days)
Population: All treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 63 | 60
Score on a scale | -1.56 (0.202) | -1.40 (0.208)

5. Secondary Outcome: Myositis Response Criteria (MRC) Total Improvement Score From Baseline to Week 24
Description: The Myositis Response Criteria (MRC) is a continuous total improvement score from baseline (range 0-100) based on the sum of the absolute percent change in the 6 core domains (weighted) used in the IMACS DOI (International Myositis Assessment and Clinical Studies definition of improvement)
  IMACS core measures are: Physician Global Assessment of Disease Activity (PGA), Patient (Subject) Global Assessment of Disease Activity (SGA), Manual Muscle Test (MMT-8), Health Assessment Questionnaire-Disability Index (HAQ-DI), Muscle Enzyme levels, Myositis Disease Activity Assessment Tool (MDAAT) Extramuscular Global Activity.
  The total improvement score ranges between 0 and 100 percent corresponds to the degree of improvement, with higher scores corresponding to a greater degree of improvement ( >/= 20 represents minimal improvement, a score of >/= 40 represents moderate improvement, and a score of >/= 60 represents major improvement).
Time Frame: From first dose to 24 weeks after first dose. (Approximately 169 days)
Population: All treated participants with both baseline and post-baseline measurements
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 62 | 58
Score on a scale | 40.83 (2.873) | 37.22 (2.963)

6. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) in the Double-Blind Period
Description: The number of treated participants experiencing an adverse event. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in participants administered a study drug and that does not necessarily have a causal relationship with the treatment.
Time Frame: From first dose up to approximately 56 days post last dose date in double-blind period or first dose in open-label period. (Up to approximately 274 days)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 73
Participants | 52 | 55

7. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAE) in the Double-Blind Period
Description: The number of treated participants experiencing a Serious Adverse Event (SAE). A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: as for outcome 6
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 73
Participants | 4 | 4

8. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) of Special Interest in the Double-Blind Period
Description: The number of treated participants experiencing adverse events of special interest: infections, malignancies, autoimmune events, local injection site reactions, and systemic injection reactions.
Time Frame: as for outcome 6
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 73
Participants
  Infections | 19 | 31
  Malignancies | 0 | 0
  Autoimmune Disorders | 2 | 3
  Systemic Injection Reactions | 4 | 5
  Local Injection Site Reactions | 1 | 0

9. Secondary Outcome: Number of Participants Experiencing Laboratory Test Abnormalities in the Double-Blind Period
Description: The number of participants experiencing laboratory test abnormalities. Laboratory analysis was performed on the following: hematology, liver and kidney function, electrolytes, other chemistry testing (glucose, protein, cardiac), and urine chemistry. Only tests with participants experiencing abnormalities were reported.
Time Frame: as for outcome 6
Population: All treated participants with at least one laboratory result for each analyte
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 73
Participants
  LOW LEUKOCYTES | 1 | 0
  HIGH LEUKOCYTES | 2 | 4
  HIGH EOSINOPHILS (ABSOLUTE) | 3 | 2
  LOW LYMPHOCYTES (ABSOLUTE) | 17 | 14
  LOW NEUTROPHILS + BANDS (ABSOLUTE) | 1 | 0
  HIGH ALANINE AMINOTRANSFERASE (ALT) | 1 | 1
  HIGH ASPARTATE AMINOTRANSFERASE (AST) | 0 | 1
  HIGH G-GLUTAMYL TRANSFERASE (GGT) | 4 | 1
  HIGH BLOOD UREA NITROGEN | 0 | 1
  HIGH CREATININE | 3 | 3
  HIGH CALCIUM, TOTAL | 1 | 0
  LOW PHOSPHORUS, INORGANIC | 0 | 1
  HIGH PHOSPHORUS, INORGANIC | 1 | 0
  HIGH SODIUM, SERUM | 0 | 1
  LOW GLUCOSE, SERUM | 4 | 3
  HIGH GLUCOSE, SERUM | 8 | 8
  HIGH PROTEIN, TOTAL | 0 | 1
  HIGH CREATINE KINASE (CK) | 0 | 4
  HIGH LACTATE DEHYDROGENASE (LD) | 0 | 1

10. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) in the Cumulative Abatacept Period
Description: as for outcome 6
Time Frame: From first dose up to approximately 56 days post last dose (up to approximately 54 months)
Population: All participants who received at least one dose of abatacept. Participants are summarized under their actual Double-Blind treatment groups, but during the Open-Label and Long-Term Extension Periods all participants received abatacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 63
Participants | 64 | 39

11. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAE) in the Cumulative Abatacept Period
Description: as for outcome 7
Time Frame: From first dose up to approximately 56 days post last dose (up to approximately 54 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 63
Participants | 14 | 8

12. Secondary Outcome: Number of Participants Experiencing Adverse Events (AE) of Special Interest in the Cumulative Abatacept Period
Description: as for outcome 8
Time Frame: From first dose up to approximately 56 days post last dose (up to approximately 54 months)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 75 | 63
Participants
  Infections and infestations | 34 | 19
  Malignancies | 0 | 0
  Autoimmune Disorders | 5 | 4
  Systemic Injection Reactions | 5 | 3
  Local Injection Site Reactions | 2 | 2

13. Secondary Outcome: Number of Participants Experiencing Laboratory Test Abnormalities in the Open-Label Period
Description: The number of participants experiencing laboratory test abnormalities. Laboratory analysis was performed on the following: hematology, liver and kidney function, electrolytes, other chemistry testing (glucose, protein, cardiac), and urine chemistry. Only tests with participants experiencing abnormalities were reported. For participants who enter the Japan open-label extension period or long-term extension period, assessments after the first dose in the open-label period and before the first dose date in the subsequent period are included. For participants who prematurely discontinue the open-label period or complete the open-label period but do not enter the Japan open-label extension period or long-term term extension period, assessments after the first dose in the open-label period and up to 56 days post last dose are included.
Time Frame: From first dose in open label period to first dose date in the subsequent period or up to 56 days post last dose (up to approximately 666 days)
Population: All participants who received at least one dose of abatacept and with at least one laboratory result for each analyte. Participants are summarized under their actual Double-Blind treatment groups, but during the Open-Label Period all participants received abatacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 69 | 63
Participants
  LOW HEMOGLOBIN | 0 | 1
  LOW LEUKOCYTES | 2 | 1
  HIGH LEUKOCYTES | 2 | 0
  HIGH EOSINOPHILS (ABSOLUTE) | 2 | 0
  LOW LYMPHOCYTES (ABSOLUTE) | 15 | 8
  HIGH LYMPHOCYTES (ABSOLUTE) | 1 | 0
  LOW NEUTROPHILS + BANDS (ABSOLUTE) | 2 | 0
  HIGH ALANINE AMINOTRANSFERASE (ALT) | 1 | 0
  HIGH ALKALINE PHOSPHATASE (ALP) | 0 | 2
  HIGH ASPARTATE AMINOTRANSFERASE (AST) | 0 | 1
  HIGH G-GLUTAMYL TRANSFERASE (GGT) | 2 | 1
  HIGH BLOOD UREA NITROGEN | 2 | 1
  HIGH CREATININE | 6 | 2
  HIGH POTASSIUM, SERUM | 1 | 0
  LOW GLUCOSE, SERUM | 1 | 1
  HIGH GLUCOSE, SERUM | 3 | 3
  LOW ALBUMIN | 0 | 1
  HIGH CREATINE KINASE (CK) | 3 | 5
  HIGH LACTATE DEHYDROGENASE (LD) | 0 | 1
  HIGH BLOOD, URINE: number analyzed (Participants) | 2 | 0
  HIGH BLOOD, URINE | 2 |
  HIGH WBC, URINE: number analyzed (Participants) | 1 | 0
  HIGH WBC, URINE | 1 |

14. Secondary Outcome: Number of Participants Experiencing Laboratory Test Abnormalities in the Long-Term Open Label Period
Description: The number of participants experiencing laboratory test abnormalities. Laboratory analysis was performed on the following: hematology, liver and kidney function, electrolytes, other chemistry testing (glucose, protein, cardiac), and urine chemistry. Only tests with participants experiencing abnormalities were reported. For participants who completed/discontinued the Long-Term Extension Period, assessments after the first dose in the Long-Term Extension Period and up to 56 days post last dose in the Long-Term Extension Period are included.
Time Frame: From first dose in the Long-Term Open Label Period up to 56 days post last dose in the Long-Term Open Label Period (up to approximately 958 days)
Population: All participants who received at least one dose of abatacept and with at least one laboratory result for each analyte. Participants are summarized under their actual Double-Blind treatment groups, but during the Long-Term Open Label Period all participants received abatacept.
Measure: Count of Participants; unit: Participants
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
Number analyzed (Participants) | 22 | 21
Participants
  LOW HEMOGLOBIN: number analyzed (Participants) | 22 | 20
  LOW HEMOGLOBIN | 1 | 0
  LOW LYMPHOCYTES (ABSOLUTE): number analyzed (Participants) | 22 | 20
  LOW LYMPHOCYTES (ABSOLUTE) | 1 | 4
  HIGH BLOOD UREA NITROGEN | 2 | 0
  HIGH CREATININE | 2 | 1
  HIGH GLUCOSE, SERUM | 1 | 0
  HIGH CREATINE KINASE (CK) | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from participants first dose to their study completion (up to approximately 55 months) SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 55 months)
Groups:
- Abatacept + Standard Treatment: Participants receive subcutaneous abatacept (125 mg weekly) in combination with standard treatment during the cumulative abatacept period.
- Placebo + Standard Treatment: Participants receive placebo (to match subcutaneous abatacept) in combination with standard treatment during the double-blind period.
Arm/Group | Abatacept + Standard Treatment | Placebo + Standard Treatment
All-Cause Mortality (participants affected / at risk) | 0/138 | 1/73
Serious Adverse Events (participants affected / at risk) | 22/138 | 5/73
Other Adverse Events (participants affected / at risk) | 31/138 | 23/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept + Standard Treatment (N=138) | Placebo + Standard Treatment (N=73)
Coronary artery disease (Cardiac disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Influenza like illness (General disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 2 | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept + Standard Treatment (N=138) | Placebo + Standard Treatment (N=73)
Influenza (Infections and infestations) | 3 | 6
Nasopharyngitis (Infections and infestations) | 9 | 8
Fall (Injury, poisoning and procedural complications) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2
Headache (Nervous system disorders) | 8 | 7
Hypertension (Vascular disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT02971683/Prot_004.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT02971683/SAP_005.pdf